CLINICAL TRIAL: NCT00197509
Title: Task Specific Training for Stroke Patients
Brief Title: Sit-to-Stand Training for Survivors of Stroke in a Long-Term Care Setting
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 04-359
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Cerebrovascular Accident
Keywords: Long-Term Care; Clinical Protocols; Sit-To-Stand
MeSH Terms: conditions — Stroke

INTERVENTIONS:
Behavioral: Sit-To-Stand Protocol and Extra Practice in Sit-To-Stand

SUMMARY:
The purpose of this study is to see if providing training using a Sit-to-Stand protocol for residents of Long-Term Care Facilities who have had a stroke will increase their independence in performing Sit-to-Stand.

DETAILED DESCRIPTION:
The implementation of a sit-to-stand protocol and extra practice has been previously validated in a rehabilitation setting, where 68% of survivors of stroke who received the training, learned to stand safely and independently from a 16" surface (the height of a regular toilet). Our findings have been supported by other research that have shown that rising from sitting is a maneuver that has been advocated for strengthening the lower extremities of elderly individuals and patients with specific disorders such as stroke. During the acute care and rehabilitation phases, considerable effort is spent to maximize a person's functional abilities following a stroke; however, continued strengthening and activity appears to stop once an individual is admitted to a LTC facility.

The main purpose of this randomized controlled trial is to examine the efficacy of implementing the Sit-to-Stand (STS) protocol with or without extra sit-to-stand practice for survivors of stroke residing in Long-Term Care (LTC) facilities on (1) their ability to learn how to stand safely and independently from a 16" surface; (2) the number of staff injuries; (3) the number of residents' falls; (4) the quality of life of the residents and staff; and (5) the translation and maintenance of knowledge of the STS protocol by staff into their daily routines.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebrovascular accident
* Reside in Long-Term Care Facility
* Have physician approval to participate in the study
* Are unable to stand up independently from a 16" surface without using their hands
* Have given informed consent

Exclusion Criteria:

* Expect to be leaving the facility in less than 24 weeks
* Have a terminal illness
* Have a total hip replacement or other orthopedic complication that prevents them from being able to safely use protocol
* Have pain that prevents their participation
* Are at higher risk for falling (i.e. blood pressure disorder/postural hypotension, vestibular disorder)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 2005-01; Study Completion 2006-02

PRIMARY OUTCOMES:
Ability to independently perform Sit-To-Stand at 12 weeks and 24 weeks
Score on quality of life measure (COOP) at 12 and 24 weeks
Score on stroke assessment (CMSA) at 12 and 24 weeks

SECONDARY OUTCOMES:
Number of resident falls at 12 and 24 weeks
Number of staff injuries at 12 and 24 weeks
Knowledge of staff on STS protocol immediately post-training, 12 and 24 weeks
Score on quality of life measure (SF-20) at 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan R Barreca, PT, BA, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton Health Sciences, Chedoke Site, Hamilton, Ontario, Canada